CLINICAL TRIAL: NCT01034865
Title: Risk Factors and Molecular Genomics for Hepatocellular Carcinoma in U.S. Patients With Chronic Liver Disease: A Case Control Study
Brief Title: Risk Factors and Molecular Genomics of U.S. Patients With Chronic Liver Disease and Hepatocellular Cancer
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Mindie H. Nguyen, Associate Professor of Medicine, Stanford University
Other Study IDs: SU-11022007-788; 76873; HEP0009 (Other: Stanford)
Record Dates: First submitted 2009-12-16; First posted 2009-12-18 (Estimated); Last update posted 2017-05-01 (Actual); Status verified 2017-04

CONDITIONS: Carcinoma, Hepatocellular
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — blood

GROUPS / COHORTS (2):
- HCC PTS: Patients with HCC with either: (i) a hepatic mass larger or equal to 5cm, or; (ii) a hepatic mass lesion confirmed by fine needle aspirate (FNA) or by pathology in the cases of surgical resection, or; (iii) a hepatic mass lesion with characteristic CT or MRI or angiographic appearance.
- LD: Patients with chronic liver disease without evidence of HCC

SUMMARY:
To identify risk factors for the development and diagnosis of hepatocellular CA in patients with chronic hepatitis C and to use the data to ultimately develop an effective screening program.

ELIGIBILITY:
Inclusion Criteria:

* For both experimental subjects and controls:

  1. Patients between older than 18 years of age of all ethnic backgrounds and genders.
  2. Patients with chronic liver disease
* For Experimental Subjects Only:

  1. Patients with HCC with a hepatic mass larger or equal to 5cm
  2. Patients with HCC with a hepatic mass lesion confirmed by fine needle aspirate (FNA) or by pathology in the cases of surgical resection
  3. Patients with HCC with a hepatic mass lesion with characteristic CT or MRI or angiographic appearance.
* For Controls Only:

Patients with chronic liver disease without evidence of HCC confirmed by either :

1. A normal AFP level

2. a negative imaging study (ultrasound, CT, or MR imaging).

3. Negative liver cancer on explants.

*Exclusion Criteria:

1. Patients who declined to participate in the study
2. Patients with a history of HIV infection
3. Patients with concurrent advanced malignancy of non-hepatic origin.
4. Patients with significant use of androgenic steroid.
5. Patients with exposure to vinyl chloride.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For Experimental Subjects Only:
  Patients with HCC
  For Controls Only:
  Patients with chronic liver disease without evidence of HCC
Sampling Method: Non-Probability Sample
Enrollment: 750 (Actual)
Dates: Start 2001-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mindie H. Nguyen, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States